CLINICAL TRIAL: NCT07134010
Title: The Impact of Perineural Injection Therapy for Adhesive Capsulitis at a Single Centre University Hospital in Selangor: A Pilot Study
Brief Title: The Impact of Perineural Injection Therapy for Adhesive Capsulitis.
Acronym: PIT; AC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Noor Hafizah Binti Samsudin Bahari, Medical Doctor, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/06/2025 (PG/FB/26)
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-06

CONDITIONS: Adhesive Capsulitis
Keywords: Perineural injection therapy in treating Adhesive Capsulitis
MeSH Terms: conditions — Bursitis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-center, two-arm, parallel-group, randomized controlled pilot trial conducted to assess the impact of Perineural Injection Therapy (PIT) on pain, shoulder mobility, and function in patients with adhesive capsulitis.
  Participants will be randomly assigned in a 1:1 ratio to either:
  Intervention Group: PIT plus conventional therapy (physiotherapy and analgesics excluding NSAIDs)
  Control Group: Conventional therapy alone (physiotherapy and analgesics including NSAIDs)
  Randomization will be implemented using a computer-generated random sequence prepared in advance and managed by an independent staff nurse not involved in treatment or outcome assessment. Allocation concealment will be ensured using sequentially numbered, opaque, sealed envelopes.
  Due to the procedural nature of PIT, blinding is not feasible for participants and treating physicians. However, outcome assessors (physiotherapists) will be blinded to group assignments to reduce bias.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Perineural injection Therapy
  Interventions: Other: perineural injection; Other: Physiotherapy
- Conventional group (Sham Comparator): Physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: perineural injection — Intervention The procedure will be performed by a rehabilitation physician who has obtained hospital-level credentialing and privileging to practice Perineural Injection Therapy (PIT). The physician has undergone hands-on training with Dr. Lyftogt-certified trainers in Malaysia.
  PIT will be administered weekly for six week (Total 6 sessions). In addition to this intervention, patient will also receive conventional therapy which is monthly outpatient physiotherapy with supplementary home-based exercise program, and oral analgesia (except NSAIDs).
  Solution: Buffered 5% dextrose.
  Pre injection: Chronic constriction injury points will be identified by palpation along the shoulder's cutaneous nerves - the suprascapular, supraclavicular, axillary, musculocutaneous, and radial nerves. These points will be marked to ensure precise targeting. Taking into account these nerve pathways, the maximum injection area for this research is set at 10 sites per session.
  Other Names: Perineural injection therapy; PIT
  Arms: Intervention group
Other: Physiotherapy — Patients will be receiving a structured home-based exercise program and will be instructed on how to perform these exercises at home. The exercise regime will be 30 minutes, 3 times a day to enhance shoulder mobility and strength in addition to the regular monthly outpatient physiotherapy session. Oral analgesics exclude NSAIDs will be prescribed as needed to manage pain.

SUMMARY:
The goal of this clinical trial is to learn if Perineural Injection Therapy (PIT) works to treat adhesive capsulitis (frozen shoulder) in adults. It will also learn about the safety of PIT.

The main questions it aims to answer are:

Does PIT reduce shoulder pain and improve shoulder range of motion more effectively than conventional therapy alone?

What side effects or medical problems do participants experience when receiving PIT?

Researchers will compare PIT to conventional therapy to see if PIT works better to treat adhesive capsulitis.

Participants will:

Receive either:

PIT once weekly for 6 weeks plus physiotherapy and oral analgesics (excluding NSAIDs), or

Conventional therapy only (physiotherapy and analgesics including NSAIDs)

Attend scheduled follow-up visits at Week 6, 1 month, and 3 months after treatment

Perform daily home-based shoulder exercises and record their analgesic use and any side effects in a patient diary

DETAILED DESCRIPTION:
Study Title:

The Impacts of Perineural Injection Therapy on Adhesive Capsulitis in a Single Centre Hospital in Selangor: A Randomized Controlled Trial Pilot Study

Study Overview :

Adhesive capsulitis, commonly known as "frozen shoulder," is a painful condition that limits shoulder movement and affects daily activities such as dressing, reaching overhead, or lifting objects. It often affects adults between the ages of 40 to 60 and can last for months or even years. For some, the condition may improve with physiotherapy and medication, but others continue to struggle with pain and stiffness.

This clinical trial aims to explore a new method of treatment called Perineural Injection Therapy (PIT). PIT involves injecting a natural sugar solution (5% dextrose) just under the skin at specific nerve areas around the shoulder. This method targets nerves that may be irritated or inflamed and helps to reduce pain and improve movement.

Although PIT has shown promising results in treating other painful conditions like nerve entrapments and joint pain, its effects on frozen shoulder have not yet been well studied. This research hopes to find out if PIT can help relieve pain, improve shoulder movement, and enhance function in people with frozen shoulder.

The current treatment options for frozen shoulder (such as physiotherapy, painkillers, and steroid injections) do not work for everyone. PIT is a non-surgical option that may help the healing process by calming nerve-related inflammation. This study will evaluate how effective PIT is and whether it is safe for use in treating adhesive capsulitis.

Participants will be randomly assigned to one of two groups:

Intervention Group: Will receive six weekly sessions of PIT combined with physiotherapy and oral pain medication (excluding NSAIDs like ibuprofen).

Control Group: Will receive only conventional therapy, including physiotherapy and standard painkillers (including NSAIDs).

All participants will:

Be evaluated for shoulder pain, range of motion, and ability to perform daily activities at the beginning of the study, at Week 6, 1-month, and 3-months after treatment.

Be taught home exercises to do daily to improve shoulder mobility and strength.

Be asked to keep a diary to record medication use and any side effects they experience.

Receive support and regular follow-ups from the research team to monitor progress and manage any issues.

Adults aged 18 and above who have been diagnosed with primary (idiopathic) adhesive capsulitis for at least 3 months and are experiencing significant shoulder pain and stiffness may be eligible. Participants must be able to understand and follow instructions in Malay or English.

People will not be eligible if they:

Have had a shoulder injection or surgery recently

Have other serious shoulder problems (like a fracture or nerve injury)

Have poorly controlled diabetes or are on certain medications that may interfere with the study

PIT is generally safe and has been used in other conditions with minimal side effects, such as mild pain or redness at the injection site. In this study, participants will be closely monitored for any adverse effects.

Potential benefits include reduced pain, improved shoulder movement, and better overall function. The information gathered may help develop better treatment options for others with frozen shoulder in the future.

Each participant will be involved in the study for approximately 3 to 4 months, including the 6-week treatment period and two follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above.
2. Diagnosed with primary adhesive capsulitis by a specialist.
3. Limitation of range of motion ≥ 50% relative to the normal side or normal reference (in patient with bilateral adhesive capsulitis) in three or more movement directions (i.e., external rotation, abduction, forward flexion, and internal rotation).
4. Chronic adhesive capsulitis shoulder pain lasting for at least 3 months.
5. Pain score of at least 4/10 on the Numerical Rating Scale (NRS) during movement, indicating at least moderate pain severity.
6. Consented to the study.

Exclusion Criteria:

1. Received any shoulder pain injection within the past 6 weeks or surgical intervention such manipulation under anesthesia, arthroscopic capsular release, or open surgery for capsular release.
2. Diagnosed with other shoulder pathology such as neurologic deficits affecting shoulder function, tumour, rotator cuff injury or fracture.
3. Has history of allergy to dextrose solution.
4. Patients receiving steroidsimmunosuppressants, psychotropic medication, or other medications that may affect, the clinical outcomes
5. Patients with haemorrhagic disease, taking anticoagulant drugs, or patients with severe diabetes mellitus having an increased risk of infection (HBA1c >8%)
6. Do not understand Malay or English language.
7. Unable to follow a 3 steps command.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | Measured at baseline (Week 0), post-treatment (Week 6), 1-month follow-up (Week 10), and 3-month follow-up (Week 18).
  Participants will rate their shoulder pain on a scale from 0 to 10, where 0 indicates "no pain" and 10 represents "worst imaginable pain."
Shoulder Range of Motion (ROM) | Measured at baseline (Week 0), post-treatment (Week 6), 1-month follow-up (Week 10), and 3-month follow-up (Week 18).
  Tool: Goniometer (standardized physical measurement)
  Passive ROM will be measured in four directions: forward flexion, abduction, internal rotation, and external rotation. Values will be recorded in degrees.

SECONDARY OUTCOMES:
Functional Outcome | Measured at baseline (Week 0), post-treatment (Week 6), 1-month follow-up (Week 10), and 3-month follow-up (Week 18).
  Tool: Shoulder Pain and Disability Index (SPADI) - validated English and Malay versions
  A self-reported questionnaire with 13 items divided into two subscales: 5 for pain and 8 for functional disability. Each item is scored from 0 (no pain/disability) to 10 (worst pain/disability), with higher scores indicating greater impairment.
Adverse Reactions | Monitored throughout the 6-week intervention
  Tool: Adverse Event Reporting Form and Patient Diary
  Description: Side effects will be classified into:
  Mild: Local pain, bruising, or redness
  Moderate: Transient numbness, swelling, or prolonged discomfort
  Severe: Infection or allergic reaction

OTHER OUTCOMES:
Frequency of Analgesic Use | Recorded weekly from baseline until the 3-month follow-up.
  Tool: Patient Diary (self-recorded)
  Description: Participants will log each use of pain medication (type and frequency) throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Noor Hafizah Samsudin Bahari, MD(UKM), Principal Investigator — Faculty of Medicine, Universiti Teknologi MARA, Sg Buloh Campus; Dr Anie Farhana Ngimron, MBBChBAO(Ireland)MRehabMed(UM), Principal Investigator — Faculty of Medicine, Universiti Teknologi MARA, Sg Buloh Campus; Assoc. Prof. Dr. Nadia Mohd Mustafah, MD(UPM), MRehabMed(UM), Principal Investigator — Faculty of Medicine, Universiti Teknologi MARA, Sg Buloh Campus
Locations (1):
- Hospital Al-Sultan Abdullah, UiTM Puncak Alam, Kuala Selangor, Selangor, Malaysia